CLINICAL TRIAL: NCT03426904
Title: Neoadjuvant Chemotherapy for Non-metastatic Locally Advanced Colon Cancer: A Prospective Multicenter Randomized Controlled Trial
Brief Title: Neoadjuvant FOLFOX Chemotherapy for Patients With Locally Advanced Colon Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Gyu-Seog Choi, Kyungpook National University Hospital, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUHCRC006
Record Dates: First submitted 2018-01-23; First posted 2018-02-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant FOLFOX (Experimental): 4 cycles of FOLFOX (Folinic acid, fluorouracil and oxaliplatin) neoadjuvant followed by surgery and 8 cycles of FOLFOX
  Interventions: Drug: Neoadjuvant FOLFOX
- Conventional adjuvant FOLFOX (Active Comparator): surgery followed by 12 cycles of FOLFOX
  Interventions: Drug: Conventional adjuvant FOLFOX

INTERVENTIONS:
Drug: Neoadjuvant FOLFOX — 4 cycles of FOLFOX neoadjuvant chemotherapy and 8 cycles of postoperative chemotherapy
  Arms: Neoadjuvant FOLFOX
Drug: Conventional adjuvant FOLFOX — 12 cycles of postoperative FOLFOX chemotherapy
  Arms: Conventional adjuvant FOLFOX

SUMMARY:
The main cause of recurrence after surgical treatment of colon cancer is distant metastasis. Neoadjuvant chemotherapy has potential benefits of improving the effectiveness of chemotherapy. Preoperative chemotherapy may eradicate microscopic metastatic cancer cells earlier than adjuvant chemotherapy, reduce cancer cell spillage during surgery, and lessen the invasiveness of surgical resection. This randomized multicenter phase III trial is assessing whether preoperative chemotherapy improves oncologic outcomes of patients with locally advanced colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed colon adenocarcinoma (> 15 cm from the anal verge)
* Radiologic T3/T4 and high risk features by CT scan
* No metastasis on CT or PET(positron emission computed tomography)
* Age ≥ 18 and ≤ 70 years
* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* No history of colorectal cancer within 5 years
* No history of chemotherapy
* Patients with childbearing potential should use effective contraception during the study and the following 6 months
* Adequate bone marrow function : white blood cell count of 2 x 109/L or more with neutrophils of1.5 x 109/L or more, platelet count of 100 x 109/L or more, hemoglobin of 9 g/dL (5,6 mmol/l) or more
* Adequate hepatobiliary function : total bilirubin of 0.4 mg/dl or less, ASAT (aspartate aminotransferase) and ALAT (alanine aminotransferase) of 2.5 x ULN (upper limits of normal) or less, Alkaline phosphatase of 1.5 x ULN or less
* Adequate renal function : GFR (Glomerular Filtration Rate) > 50ml/min by Wright or Cockcroft formula
* Signed written informed consent obtained prior to any study specific screening procedures

Exclusion Criteria:

* Age > 70 years and < 18 years
* Rectal cancer : 15 cm or less from the anal verge
* Complicated colon cancer (complete obstruction, perforation, bleeding)
* Metastatic colon cancer
* Known hypersensitivity reaction to any of the components of study treatments
* Inflammatory bowel disease
* Hereditary nonpolyposis colorectal cancerHNPCC, familial Adenomatous Polyposis
* Clinically relevant coronary artery disease or history of myocardial infarction in the last 6 months, high risk of uncontrolled arrhythmia
* Galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Pregnancy or breast-feeding period
* Serious non-healing wound or bone fracture
* Medical, geographical, sociological, psychological or legal conditions that would not permit the patient to complete the study or sign informed consent
* Any significant disease which, in the investigator's opinion, would exclude the patient from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2028-12-28 (Estimated); Study Completion 2031-12-28 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival after randomization | 3 years after randomization

SECONDARY OUTCOMES:
Overall survival | 3 year after randomization
Radiological assessment of response to neoadjuvant treatment | 6 months after surgery
Pathological assessment of response to neoadjuvant treatment | 1 months after surgery
  Replacement of the tumor by fibrous or fibro-inflammatory granulation tissue
Surgical complication | 60 days after surgery
Length of hospital stay | 60 days after surgery
Quality of life (EORTC QLQ-C30) | before treatment, before surgery, 3 months after surgery, 6 months after surgery, 1 year after surgery
  QLQ (quality of life questionnaire)
Quality of life (EORTC QLQ-C38) | before treatment, before surgery, 3 months after surgery, 6 months after surgery, 1 year after surgery
Toxicity of chemotherapy | 1 year
  Toxicity : incidence of chemotherapy-related adverse events according to CTCAE (Common Terminology Criteria for Adverse Events) v4.0
Incidence of completion of chemotherapy | 1 year
Accuracy of CT staging | 1 year
Total cycles of perioperative chemotherapy | 1 year
Pathological tumor stage | 1 month after surgery
  Colon cancer stage by AJCC 8th edition

CONTACTS AND LOCATIONS:
Overall Officials: Soo Yeun Park, MD, Study Director — Kyungpook National University Chilgok Hospital; Gyu-Seog Choi, MD, PhD, Principal Investigator — Kyungpook National University Chilgok Hospital
Locations (4):
- South Korea (4):
  - Chonnam National University Hwasun Hospital, Hwasun, Chonnam
  - Kyungpook National University Chilgok Hospital, Daegu
  - Asan Medical Center, Seoul
  - The Catholic Univ. of Korea St. Vincent's Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No